CLINICAL TRIAL: NCT04118270
Title: Shared Decision-Making: Implementing the AFib 2getherTM Mobile App
Brief Title: Shared Decision-Making: AFib 2gether Mobile App
Acronym: AFib 2gether
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Alok Kapoor, Associate Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: H00018053
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation New Onset

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- AFib 2gether(TM) App (Experimental): Patients with known Atrial Fibrillation will be assigned to download and use an app targeted at determining stroke risk and increasing knowledge of Atrial Fibrillation and stroke risk along with treatment options and will use this information to facilitate a discussion with their cardiovascular provider.
  Interventions: Device: Afib 2gether TM Mobile Application

INTERVENTIONS:
Device: Afib 2gether TM Mobile Application — The Afib 2gether mobile app determines a patient's stroke risk through a series of questions that the patient will answer in the app.

SUMMARY:
Shared Decision-Making: AFib 2gether™ is a research study that focuses on a mobile application developed by Pfizer, Inc with consultation from Dr McManus' called AFib 2gether™. Through this app, patients can determine their risk of stroke due to atrial fibrillation and prioritize questions and concerns for discussion with their cardiology provider.

ELIGIBILITY:
Inclusion Criteria:

Providers:

* Caring for at least 3 patients aged 18 years and older
* Have at least 3 patients with International Classification of Diseases tenth revision (ICD-10) diagnostic code consistent with atrial fibrillation (AF) or atrial flutter
* Have at least 3 patients with a CHA2DS2-VASc stroke risk score of 2 or more
* Have at least 3 patients who are not on anticoagulation
* Have at least 3 patients with upcoming appointments within the next 4 months

Patients:

* Age 18+
* Preferred language is English
* Atrial fibrillation diagnosis
* Chads vasc score 2 or higher
* Not on anticoagulants
* No watchman or atrial appendage closure
* Had an ambulatory care center (ACC) cardiology appointment in the past 12 months
* Future appointment in the next 4 months with the same provider

Exclusion Criteria:

Providers:

* Providers who do not care for at least 3 patients aged 18 years and older
* Have patients that do not have an ICD-10 diagnostic code consistent with AF or atrial flutter
* Does not have patients with a CHA2DS2-VASc stroke risk score of 2 or more
* Their patients are on anticoagulation
* Their 3 patients do not have an upcoming visit within the next 4 months

Patients:

* Under the age of 18; patients
* No ICD-10 diagnostic code consistent with AF or atrial flutter
* Did not have a visit with a cardiovascular medicine specialist in the previous one year
* Patients with a CHA2DS2-VASc score less than 2
* Currently prescribed an anticoagulant
* No upcoming cardiology visit in the next 3 months
* Has a WATCHMAN device or left atrial appendage closure surgery
* On hospice or for whom life expectancy is less than six months and patients
* Bleeding episode or fall with injury in the last four weeks
* Does not speak English
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alok Kapoor, MD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapoor A, Hayes A, Patel J, Patel H, Andrade A, Mazor K, Possidente C, Nolen K, Hegeman-Dingle R, McManus D. Usability and Perceived Usefulness of the AFib 2gether Mobile App in a Clinical Setting: Single-Arm Intervention Study. JMIR Cardio. 2021 Nov 19;5(2):e27016. doi: 10.2196/27016. PMID 34806997
- [Derived] Kapoor A, Andrade A, Hayes A, Mazor K, Possidente C, Nolen K, Hegeman-Dingle R, McManus D. Usability, Perceived Usefulness, and Shared Decision-Making Features of the AFib 2gether Mobile App: Protocol for a Single-Arm Intervention Study. JMIR Res Protoc. 2021 Feb 24;10(2):e21986. doi: 10.2196/21986. PMID 33625361

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We identified 40 patients seeing 13 cardiology providers. Of the 40 patients, 2 were later found ineligible and 1 patient was disenrolled due to provider preference leaving us with 37 patient encounters to analyze. Of the 13 providers, 10 completed the accuracy assessment.
Groups:
- Providers: Providers caring for the patients with known Atrial Fibrillation will be asked to review the patients' stroke risk score on the AFib 2gether app and compare to their clinical assessment for accuracy.
Period: Overall Study
Arm/Group | AFib 2gether(TM) App | Providers
Started | 37 | 13
Completed Provider Accuracy Assessment | 0 (Only the Providers were eligible for completing the Provider Accuracy Assessment.) | 10
Completed | 37 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Information about patient characteristics (such as demographics) was collected in addition to the patients stroke risk score and reason why they were not on an anticoagulant (AC) prior to their appointment in the cardiology clinic. Baseline data for providers such as provider characteristics was not collected.
Groups:
- Providers: Providers caring for the patients with known Atrial Fibrillation will be asked to review the patients' stroke risk score on the AFib 2gether app and compare to their clinical assessment for accuracy. Baseline measures were not collected for providers.
- Total: Total of all reporting groups
Arm/Group | AFib 2gether(TM) App | Providers | Total
Number analyzed (Participants) | 37 | 0 | 37
Age, Customized [Count of Participants; unit: Participants] — The patients age was collected through the Electronic Medical record (EHR).
  Participants
    Age: 75+ | 17 |  | 17
    Age: 65-74 | 14 |  | 14
    Age: <65 | 6 |  | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 |  | 11
  Male | 26 |  | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 36 |  | 36
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Stroke Risk Score [Count of Participants; unit: Participants] — The CHA2DS2-VASc scale is an evaluation of stroke risk in patients with atrial fibrillation. The scale is a composite of 7 questions (based on age, sex, congestive heart failure history, hypertension history, stroke/transient ischemic attack/thromboembolism history, vascular disease history, diabetes history), with an overall scale score of 0 to 9, with low scores indicating low risk for stroke, and high scores indicating high risk for stroke.
  Participants
    CHA2DS2-VASc score: 2 | 9 |  | 9
    CHA2DS2-VASc score: 3 | 10 |  | 10
    CHA2DS2-VASc score: 4 | 9 |  | 9
    CHA2DS2-VASc score: 5 | 6 |  | 6
    CHA2DS2-VASc score: 6 | 2 |  | 2
    CHA2DS2-VASc score: 7 | 0 |  | 0
    CHA2DS2-VASc score: 8 | 0 |  | 0
    CHA2DS2-VASc score: 9 | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient MARS Scores
Description: Patients evaluated the perceived usefulness of the AFib 2gether mobile application by taking the Mobile App Rating Scale (MARS) questionnaire. This evaluated 3 domains: functionality, aesthetics, and a star-based question. These scores are rated 1-5 with 5 being the highest (best) score.
Time Frame: Immediately after visit
Population: Patients with a stroke risk score of 2 or higher and have a diagnosis of AF.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patient: Patients with a stroke risk score of 2 or higher and have a active diagnosis of atrial fibrillation (AF).
Arm/Group | Patient
Number analyzed (Participants) | 37
score on a scale
  Functionality | 4.51 (0.61)
  Aesthetics | 4.26 (0.51)
  Star-Based | 4.24 (0.89)

2. Secondary Outcome: Provider MARS Scores
Description: Providers were asked to navigate the app features and rate their overall opinion of the mobile app by answering questions using the Mobile App Rating Scale (MARS). This scale evaluates 3 domains: functionality, aesthetics, and a star-based rating question. These scores are rated 1-5 with 5 being the highest (best) score.
Time Frame: Immediately after visit.
Population: Providers are considered to be enrolled in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Provider: Providers who are caring for patients who have a stroke risk of 2 or higher and have an active AF diagnosis.
Arm/Group | Provider
Number analyzed (Participants) | 13
units on a scale
  Functionality | 4.19 (0.50)
  Aesthetics | 4.04 (0.50)
  Star-Based | 3.76 (0.44)

3. Secondary Outcome: Reason Why the Patient Was Not on AC Prior to Their Appointment
Description: This was an evaluation of why the patient was not on an anticoagulant (AC) prior to their appointment.
Time Frame: Immediately after visit
Measure: Number; unit: participants
Groups:
- Patient: Patients with a stroke risk score of 2 or greater and an active diagnosis of AF.
Arm/Group | Patient
Number analyzed (Participants) | 37
participants
  Low AF Burden | 16
  Refused | 10
  Not Listed | 5
  Fall Risk | 1
  GI Bleed | 2
  Other Bleed | 3

4. Other Pre Specified Outcome: Number of Patients Placed on Anticoagulation After Cardiology Appointment
Description: This outcome measures the number of patient participants with a CHA2DS2-VASc stroke scale score of 2 or higher who are placed on anticoagulation therapy following cardiology appointment. Patients switch to AC will be monitored via the electronic health record. The CHA2DS2-VASc scale is an evaluation of stroke risk for patients with atrial fibrillation. The scale is a composite of 7 questions, with an overall scale score of 0 to 9, with low scores indicating low risk for stroke, and high scores indicating high risk for stroke.
Time Frame: up to 6 months
Population: Patients with AF with a stroke risk score that is 2 or higher.
Measure: Count of Participants; unit: Participants
Arm/Group | AFib 2gether(TM) App
Number analyzed (Participants) | 37
Participants | 12

5. Secondary Outcome: Afib 2gether Accuracy Assessment
Description: The provider was asked to review the patients stroke risk score on the AFib 2gether app and compare to provider clinical assessment for accuracy. The number of accurate scores were recorded. Ten of the original thirteen providers completed this assessment.
Time Frame: Immediately after visit.
Population: Providers are considered enrolled in the study.
Measure: Number; unit: accurate scores
Arm/Group | Provider
Number analyzed (Participants) | 10
accurate scores | 10

ADVERSE EVENTS:
Time Frame: The proposed study involves no more than minimal risk to participants but adverse events can be self reported by participants for the duration of the study, 6 months.
Arm/Group | AFib 2gether(TM) App | Providers
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/13
Other Adverse Events (participants affected / at risk) | 0/37 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT04118270/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT04118270/SAP_002.pdf